CLINICAL TRIAL: NCT03012139
Title: Cancer-Associated Muscle Atrophy and Weakness: An Investigation of Etiology
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rajiv Kumar, M.D., PI, Mayo Clinic
Other Study IDs: 16-007030
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Cancer; Cachexia; Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Cachexia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, and skeletal muscle tissue will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cancer with cachexia: Men and women (ages 35-80 years) with cancer cachexia (≥5% drop in body mass in less than 12 months)
- Cancer without cachexia: Men and women (ages 35-80 years) with cancer but without cachexia of similar age and sex as the group with cachexia
- No cancer: Men and women (ages 35-80 years) without cancer, but similar age and sex as groups with cancer.

SUMMARY:
This study is designed to gain a better understanding of the mechanisms leading to muscle wasting and metabolic abnormalities in skeletal muscle of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-80 years
* Diagnosis of metastatic cancer with cachexia (≥5% drop in body mass in less than 12 months), metastatic cancer without cachexia (<5% drop in body mass in 12 months) or no history of cancer but similar in age and sex as other groups.

Exclusion Criteria:

* Current use of vitamin D analogs
* Fasting plasma glucose ≥126 mg/dL
* Renal failure (serum creatinine > 1.5mg/dl)
* Chronic active liver disease (Bilirubin > 17mmol/L, AST>144IU/L, or ALT>165IU/L)
* Contraindications to MRI (e.g., pacemaker, ferrous materials within body).
* Active coronary artery disease or history of unstable macrovascular disease (unstable angina, myocardial infarction, stroke, and revascularization of coronary, peripheral or carotid artery within 3 months of recruitment)
* Renal insufficiency/failure (serum creatinine > 1.5mg/dl)
* Oral warfarin group medications or history of blood clotting disorders.
* People who have taken Bevacizumab
* Platelet count <100,000 per uL
* Pregnancy or breastfeeding
* Alcohol consumption greater than 2 glasses/day or other substance abuse
* Untreated or uncontrolled thyroid disorders
* Debilitating chronic disease (at the discretion of the investigators)
* Previous injury/trauma/surgery to the region being measured without full recovery
* Pain in the area to be assessed
* Any medical condition affecting the ability to execute a maximal muscle contraction
* The presence of infections, highly communicable diseases (AIDS, active tuberculosis, veneral disease, hepatitis) or metastatic bone disease that may interfere with safely executing maximal effort.
* Significant neurological or musculoskeletal disorders or disease that may interfere with safely executing maximal contraction
* Any congenital, developmental, or other bone disease or previous surgeries that may interfere with successful testing

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit patients with metastatic cancer with or without evidence of cachexia, defined as ≥5% drop in body mass in less than 12 months. Controls without cancer but similar in age, sex, and body mass index will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-01; Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle oxidative capacity | Approximately within a month of recruitment
  Muscle oxidative capacity will be measured by magnetic resonance spectroscopy
Skeletal muscle protein synthesis | Approximately within a month of recruitment
  Muscle protein synthesis will be measured in the postabsorptive state from the rate of incorporation of isotopically labeled amino acids given intravenously.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Kumar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided